CLINICAL TRIAL: NCT04603755
Title: Electrical Impedance Tomography: Collapse in Dependent Areas as a Predictor of Response to Prone Position Ventilation in COVID-19 Acute Respiratory Distress Syndrome
Acronym: COVIDEIT
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-16; 2020-A02823-36 (Other: IDRCB)
Record Dates: First submitted 2020-10-24; First posted 2020-10-27 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV Infection; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrical Impedance tomography — Electrical Impedance tomography recording during 5 minutes every day during 7 days

SUMMARY:
There are several clinical presentations of SARS-CoV-2 infection. Among the severe forms, pulmonary involvement with respiratory failure is common. Although severe lung involvement with SARS-CoV-2 meets the Berlin criteria for Acute Respiratory Distress Syndrome (ARDS), it differs from classic ARDS in that compliance (reflecting distensibility of the lung parenchyma) is frequently preserved.

If the interest of Electrical Impedance Tomography has been demonstrated in classical ARDS, this is not the case in ARDS with COVID-19.

However, the use of this technique in this particular patient population would make it possible to distinguish patients with severe hypoxemia linked to derecruitment from those without derecruitment, in whom hypoxemia is more likely to be linked to the loss of hypoxic vasoconstriction.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit for SARS-CoV-2 ARDS
* Under controlled invasive ventilation for less than 7 days

Exclusion Criteria:

* Pneumothorax
* Deformation of the rib cage
* Contraindication to Electrical Impedance Tomography
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is composed of patients who have been admitted to the intensive care unit for SARS-CoV-2 ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Coefficient of correlation between the percentage of derecruitment of dependent areas (measured with Electrical Impedance Tomography) and the response to prone position | Up to 7 days
  The percentage of derecruitment of dependent areas will be measured every day with Electrical Impedance Tomography.
  The response to prone position will be assessed every day.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital de la Timone, Marseille
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cardinale M, Boussen S, Cungi PJ, Esnault P, Mathais Q, Bordes J, Meaudre E, Goutorbe P. Lung-Dependent Areas Collapse, Monitored by Electrical Impedance Tomography, May Predict the Oxygenation Response to Prone Ventilation in COVID-19 Acute Respiratory Distress Syndrome. Crit Care Med. 2022 Jul 1;50(7):1093-1102. doi: 10.1097/CCM.0000000000005487. Epub 2022 Feb 11. PMID 35200196